CLINICAL TRIAL: NCT04690101
Title: Treatment of Choledocolithiasis by Laparoscopic Exploration of The Bile Tract After Failed Endoscopic Cholangiopancreatography
Brief Title: Treatment of Choledocolithiasis by Laparoscopic Exploration
Status: Completed | Type: Observational
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Israel De Alba Cruz, Principal Investigator, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Other Study IDs: IDC001
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: none, this is an observational study — none, this is an observational study

SUMMARY:
There are three treatment options for choledocholithiasis: endoscopic retrograde cholangiopancreatography (ERCP) followed by laparoscopic cholecystectomy; laparoscopic exploration of the main bile duct with concomitant cholecystectomy; and open cholecystectomy with exploration of the main bile duct. A retrospective, descriptive, observational study was taken of patients with a diagnosis of cholecystocholedocholithiasis that failed ERCP and who underwent laparoscopic cholecystectomy with exploration of the bile duct.

DETAILED DESCRIPTION:
this study was revision of clinical files.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cholecyto-choledocholithiasis with failed ERCP and who were taken to LCDE in the General Surgery service

Exclusion Criteria:

* Less than 18 year old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of cholecyto-choledocholithiasis with failed ERCP and who were taken to LCDE in the General Surgery service of the General Ignacio Zaragoza
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-01-31 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
TREATMENT OF CHOLEDOCOLITHIASIS | 2009-2018
  TREATMENT OF CHOLEDOCOLITHIASIS AFTER FAILED ENDOSCOPIC CHOLANGIOPANCREATOGRAPHY

IPD SHARING:
Plan to Share IPD: Undecided